CLINICAL TRIAL: NCT04950296
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study of the Efficacy and Safety of L. Plantarum UALp-05TM in Diarrhea- Predominant-irritable Bowel Syndrome
Brief Title: To Study the Efficacy and Safety of L. Plantarum UALp-05TM in Diarrhea- Predominant-irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UAS201003/LPLANTARUMUALP05IBS
Record Dates: First submitted 2021-06-16; First posted 2021-07-06 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-01

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — Exercise; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: L. plantarum UALp-05TM, (Active Comparator): One capsule to be taken orally before lunch with a glass of water. In case the dose is missed, advise participant to take before dinner.
  Interventions: Other: Group I: L. plantarum UALp-05TM,
- Group II: L. plantarum UALp-05TM, (Active Comparator): One capsule to be taken orally before lunch with a glass of water. In case the dose is missed, advise participant to take before dinner.
  Interventions: Other: Group II: L. plantarum UALp-05TM,
- Microcrystalline Cellulose (Placebo Comparator): One capsule to be taken orally before lunch with a glass of water. In case the dose is missed, advise participant to take before dinner.
  Interventions: Other: Microcrystalline cellulose

INTERVENTIONS:
Other: Group I: L. plantarum UALp-05TM, — One capsule to be taken orally before lunch with a glass of water. In case the dose is missed, advise participant to take before dinner.
  Other Names: Active
  Arms: Group I: L. plantarum UALp-05TM,
Other: Group II: L. plantarum UALp-05TM, — One capsule to be taken orally before lunch with a glass of water. In case the dose is missed, advise participant to take before dinner.
  Other Names: Active
  Arms: Group II: L. plantarum UALp-05TM,
Other: Microcrystalline cellulose — One capsule to be taken orally before lunch with a glass of water. In case the dose is missed, advise participant to take before dinner.
  Other Names: Placebo
  Arms: Microcrystalline Cellulose

SUMMARY:
Several probiotic strains have shown beneficial outcomes in IBS patients, particularly among the Lactobacillus and Bifidobacterium genera, Lactobacillus plantarum (recently reclassified as Lactiplantibacillus plantarum) is a frequently isolated species of the healthy human GI tract that has been studied in numerous GI clinical studies, including for IBS.In the present study, the efficacy and tolerability of L. plantarum (UALp-05TM), will be evaluated in individuals with IBS-D.

DETAILED DESCRIPTION:
Several strains of Lactobacillus genus have previously been assessed in patients with IBS in multiple randomized controlled trials, demonstrating the efficacy of these strains in reducing IBS-related symptoms such as abdominal pain, distension and flatulence. We hypothesize the L. plantarum UALp-05 strain to benefit research participants by reducing pain severity, normalizing diarrhea predominant stool type and subsequently improving quality of life (QOL) standards. The current study with L. plantarum UALp-05, will include a lower dose of 1 billion CFU/day (considered a low dose among probiotic IBS studies) and a higher dose of 10 billion CFU/ day (considered a mid-point dose among probiotic IBS studies) for a period of 8-weeks.Each probiotic dosage group will be assessed individually in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 70 years.
2. Participants with Irritable bowel syndrome (IBS) as per Rome IV IBS criteria:

   Recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria:
   * Related to defecation (Maybe increased or decreased by defecation)
   * Associated with a change in the frequency of stool (increase in frequency)
   * Associated with a change in the form (appearance) of stool
3. History of abnormal bowel movements, which are predominantly diarrhea (more than one-fourth (25%) of bowel movements with BSS Types 6-7 and less than one-fourth (25%) with BSS Types 1-2) in the last one month prior to screening.
4. Average APS-NRS score of ≥ 6 for last 3 months prior to screening visit.
5. Fasting blood glucose levels ≤ 125 mg/dL (6.94 mmol/l).
6. Hemoglobin ≥ 10 g/dL.
7. Able to comply and perform the procedures requested by the protocol (consumption of study medications, filling scheduled eDiary for health updates, biological sample collection procedures and study visit schedule).
8. Participants with access to western toilet facilities.
9. Participants with non-vegetarian dietary preferences (Note: Non-vegetarian food will be defined as food derived from animals, birds, fish, shell-fish, etc)
10. Participants consuming non-vegetarian food for at least 2 times in a week.
11. SpO2 ≥ 96% as assessed by fingertip pulse oximetry
12. Participants who are sufficiently literate to understand the essence of the study, are informed about the purpose of the study, and understand their rights.
13. Participants who are able to give written informed consent and are willing to participate in the study.

Exclusion Criteria:

1. Participants not meeting IBS-D diagnostic criteria (i.e. IBS-Constipation, Mixed or Unclassified).
2. Uncontrolled abnormal Thyroid Stimulating Hormone (TSH) value which is < 0.35 or > 4.94 μIU/mL.
3. Uncontrolled Type II DM (Controlled Type II diabetics can be included upon investigator's discretion).
4. Type I diabetes.
5. Uncontrolled hypertension defined as SBP ≥ 140 mm Hg and/or DBP ≥ 90 mm Hg.
6. Use of probiotics and/or prebiotics (In the form of supplements) within the last 4 weeks prior to screening.
7. Use of medicines (Prescription, OTC, etc), health supplements or herbal medicines expected to promote gut health and alleviate IBS related complications within the last four 4 months prior to screening.
8. Established diagnosis of Helicobacter pylori infection in last 3 months prior to screening.
9. History of surgical resection of the stomach, small intestine or large intestine.
10. Participants with acute gastroenteritis.
11. History or complications of inflammatory bowel disease (Crohn's disease or ulcerative colitis) or ischemic colitis.
12. Participants with complications from infectious enteritis.
13. History of any diet-based intolerance (gluten or lactose intolerance).
14. History of or complications from malignant tumors.
15. History of any significant neurological or psychiatric condition which may affect study participation or inference of study outcomes.
16. Consumption of psychotropic agents in the last 1 year prior to screening.
17. History (in past 2 years) of smoking or currently smoking or using any form of smokeless tobacco.
18. Participation in other clinical trials in last 90 days prior to screening.
19. Participants with heavy alcohol consumption, defined as:

    * For men: More than 14 standard alcoholic drinks (SAD)/week or more than 4 SAD in a day.
    * For women: More than 7 SAD/week or more than 3 SAD in a day. (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol).
20. Participants who have a clinically active state of systemic illness, which may include but is not limited to cardiovascular, endocrine, immune, respiratory, hepatobiliary, kidney and genitourinary, neuropsychiatric, and gastrointestinal system. To be ruled out by physician based on prior history and physical examination.
21. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
22. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale | Day 0, Day 56
  To evaluate the effect of IP consumption on change in Irritable Bowel Syndrome Symptom Severity Scale total score on day 56 from baseline (Day 0) in comparison to placebo.
  A score on a scale, include 0 to 100 pointer scale the minimum score is the better outcome and maximum values is worse outcome.

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale | Day 28
  To evaluate the effect of Investigational Product on global assessment of Irritable Bowel Syndrome symptoms, as assessed by the change in Irritable Bowel Syndrome Symptom Severity Scale total score on day 28 from baseline (day 0) in comparison to placebo. A score on a scale, include 0 to 100 pointer scale the minimum score is the better outcome and maximum values is worse outcome.
Abdominal Pain Severity Numeric Rating Scale | Screening, Day 0, Day 28 and Day 56
  To evaluate the effect of IP on abdominal pain severity (11-point scale), as assessed by the change in Abdominal Pain Severity Numeric Rating Scale score on day 56 from baseline (day 0) in comparison to placebo. A score on a scale, include 0 to 10 pointer scale the minimum score is the better outcome and maximum values is worse outcome.
Bristol Stool Scale | Screening, Day 0, Day 28 and Day 56
  To evaluate the effect of IP on percentage of study population achieving normal stool consistency, as assessed by Bristol Stool Scale on day 56 from baseline (day 0) in comparison to placebo. Bristol Stool Scale (BSS), a validated ordinal scale of stool types ranging from 1 through 7, with types 1-2 and 6-7, in conjunction with other symptoms, indicative of constipation and diarrhea, respectively. Types 3-5 are generally considered to be the most normal stool form and are the modal stool forms in cross-sectional surveys of healthy adults.
Irritable Bowel Syndrome Symptom Severity Scale percent responder | Day 56
  To evaluate the effect of IP on percent responders defined by clinically significant Irritable Bowel Syndrome Symptom Severity Scale total score improvement on day 56 in comparison to placebo.
  A score on a scale, include 0 to 100 pointer scale the minimum score is the better outcome and maximum values is worse outcome.
Irritable Bowel Syndrome -Quality of Life | Day 0, Day 28 and Day 56
  To evaluate the effect of IP on quality of life as assessed by the change in Irritable Bowel Syndrome -Quality of Life score on day 56 from baseline (day 0) in comparison to placebo.
  34 set of Questionnaire indication following score 1=Not at all, 2=Slightly, 3=Moderately, 4=Quite a bit, 5=A great deal, the minimum score is the better outcome and maximum values is worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramesh Dargad, Principal Investigator — Stress test clinic
Locations (12):
- India (12):
  - Apex Gastro Clinic and Hospital,, Ahmedabad, Gujarat
  - SN Gastro and Liver Clinic, Ahmedabad, Gujarat
  - Ahmedabad Gastro Associates,, Ahmedabad, Gujarat
  - Aman Hospital and research center, Vadodara, Gujarat
  - My Health Clinic,, Mumbai, Maharashtra
  - Dr. Khanna Clinic,, Mumbai, Maharashtra
  - Stress Test Clinic, Mumbai, Maharashtra
  - Samarth Digestive Disease Centre, Mumbai, Maharashtra
  - Rahate Surgical Hospital,, Nagpur, Maharashtra
  - Ashirwad Hospital And Research Centre,, Ulhasnagar, Maharashtra
  - Shubham Sudbhawana Superspeciality Hospital,, Varanasi, Uttar Pradesh
  - Khannas Clinic, Varanasi, Uttar Pradesh